CLINICAL TRIAL: NCT05924373
Title: A Phase 2, Randomized, Double-blind, Parallel, Placebo-controlled Study to Evaluate Efficacy and Safety of Local Injection of Human Dental Pulp Mesenchymal Stem Cells for the Treatment of Chronic Periodontitis Patients.
Brief Title: Human Dental Pulp Mesenchymal Stem Cells for the Treatment of Chronic Periodontitis Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Capital Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH-hDP-MSC-102
Record Dates: First submitted 2023-05-17; First posted 2023-06-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2023-05

CONDITIONS: Periodontitis
Keywords: Human Dental Pulp Stem Cell
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, double-blind, parallel, placebo-controlled study
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- single-dose group (Experimental): Human Dental Fulp Stem Cells Injection: 1X 10^7 cells/periodontaldefect site.
  Interventions: Drug: Human Dental Fulp Stem Cells
- two-dose group (low-dose) (Experimental): Human Dental Pulp Stem Cells Injection: 1X 10^6 cells/periodontaldefect site. Continuous administration twice, with an interval of 89 days between each administration.
  Interventions: Drug: Human Dental Fulp Stem Cells
- two-dose group (high-dose) (Experimental): Human Dental Pulp Stem Cells Injection: 1X 10^7 cells/periodontaldefect site. Continuous administration twice, with an interval of 89 days between each administration.
  Interventions: Drug: Human Dental Fulp Stem Cells

INTERVENTIONS:
Drug: Human Dental Fulp Stem Cells — Investigational drugs: Based on the initial periodontal treatment (supragingival cleansing, subgingival scaling and root planning), human pulp stem cell injections will be given for a single or two local injection
  Other Names: Initial periodontal therapy

SUMMARY:
The primary objective:To evaluate the efficacy of different administration protocols of human dental pulp mesenchymal stem cells for the treatment of chronic periodontitis patients.

The secondary objective:To evaluate the safety of different administration protocols of human dental pulp mesenchymal stem cells for the treatment of chronic periodontitis patients.

The exploratory objective:To investigate the effects of human dental pulp mesenchymal stem cells on biomarkers in gingival crevicular fluid in chronic periodontitis patients.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel, placebo-controlled study, including three treatment groups which are single-dose group, two-dose group (low-dose), and two-dose group (high-dose). The patients of single-dose group will receive only one dose on day 1 (D1), and the patients of two-dose groups will receive one dose on D1 and D90 respectively. 68 participants will be enrolled in each group, and be randomized (3:1) to receive human dental pulp mesenchymal stem cells (hDP-MSCs) or placebo (normal saline). Participants in the single-dose group and the two-dose group (high-dose) will receive local injection of 1.0 × 107 hDP-MSCs (0.6mL normal saline suspension) / periodontal defect site or 0.6mL normal saline / periodontal defect site, and participants in the two-dose group (low-dose) will receive local injection of 1.0 × 106 hDP-MSCs (0.6mL normal saline suspension) / periodontal defect site or 0.6mL normal saline / periodontal defect site. All participants will receive basic periodontal treatment simultaneously.

Dosing interval: the dosing interval is set at 89 days, which is based on the results of preclinical trials of hDP-MSCs, the improvement of periodontitis observed on D90 after hDP-MSCs administration, and good safety profile in phase 1 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible to be included in the study only if all of the following criteria apply:

1)18 to 65 years old (including threshold), unlimited gender; 2)Radiological examination of the periodontal defect site shows angular bone defect; 3)The probing depth (PD) at the periodontal defect site is 4 to 8 mm at baseline; 4)Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures; 5)Voluntarily participate in the clinical study, understand and sign the informed consent;

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:

  1. Participants with severe periodontal diseases (alveolar bone resorption exceeds two-thirds of the tooth root length) which affect the investigator's judgment;
  2. The grade of studied tooth looseness ≥ grade 3 at baseline (only buccolingual movement is defined as grade 1; buccolingual and mesiodistal movement is grade 2; vertical loosening is grade 3);
  3. The studied tooth with occlusal trauma which affect the investigator's judgment;
  4. Participants with surgical treatment of previous periodontal defect sites and adjacent periodontal tissues;
  5. Participants with non-steroid anti-inflammatory drug, steroid hormone therapy, and/or other hormone (except topical hormones) treatment within past 3 months of the screening visit, and/or previous use of bisphosphonates;
  6. Participants with severe systemic infection within past 3 months of the screening visit, or antibiotics treatment within past 72h of the screening visit;
  7. Participants with uncontrolled hypertension within 1 month before screening (defined as sitting systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg after receiving the optimal antihypertensive therapy);
  8. Participants with severe or uncontrolled diseases in any system (cardiac, hepatic, renal, respiratory, hematologic, endocrine, nervous, or psychiatric);
  9. Participants are known to be allergic to any materials that may be used during surgery (allergy-prone constitution or history of allergy to blood products);
  10. Any of the following abnormalities in clinical laboratory tests at screening: ALT > 3 ULN, total bilirubin > 1.5 ULN, serum creatinine > 1.5 ULN, international normalized ratio (INR) ≥ 1.5 ULN or activated partial thromboplastin time (APTT) ≥ 1.5 ULN (except for patients receiving anticoagulation therapy), Hb < 80 g/L, or PLT < 75.0×109/L;
  11. Positive result for any of the following tests at screening: hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab), or Treponema pallidum antibody (TP-Ab);
  12. Females who are pregnant or breastfeeding;
  13. Participants and their partners who plan to conceive or do not agree to use the effective non-pharmacological method of contraceptive during the trial from screening visit to 6 months after the end of the trial;
  14. Participants participated in other clinical studies within past 3 months of the screening visit;
  15. Participants with a history of smoking addiction within past 12 months of the screening visit (the number of cigarettes smoked per day ≥ 10); Other circumstances deemed inappropriate by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-03-07 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in height of the periodontal bone defect | at baseline, 90 days, 180 days
  Changes from baseline in height of the periodontal bone defect which will be examined by CBCT at D90±7 and D180±14 (primary efficacy endpoint)

SECONDARY OUTCOMES:
Changes from baseline in respiration rate of Vital Signs | within 180 days after administration
  Respiratory rate, in beats per minute
Changes from baseline in heart rate of Vital Signs | within 180 days after administration
  Heart rate in beats per minute
Changes from baseline in blood pressure of Vital Signs | within 180 days after administration
  Blood pressure in mmHg, both systolic and diastolic blood pressure will be measured.
Changes from baseline in body temperature of Vital Signs | within 180 days after administration
  Body temperature in Celsius degree
Changes from baseline in red blood cell count of Laboratory Examination | within 180 days after administration
  Red blood cell count in whole blood is reported in the form of number
Changes from baseline in white blood cell count of Laboratory Examination | within 180 days after administration
  White blood cell count in whole blood is reported in the form of number
Changes from baseline in neutrophil count of Laboratory Examination | within 180 days after administration
  Neutrophil count in whole blood is reported in the form of number
Changes from baseline in lymphocyte count of Laboratory Examination | within 180 days after administration
  Lymphocyte count in whole blood is reported in the form of number
Changes from baseline in platelet count of Laboratory Examination | within 180 days after administration
  Platelet count in whole blood is reported in the form of number
Changes from baseline in hemoglobin of Laboratory Examination | within 180 days after administration
  Changes of hemoglobin concentration（g/dL）in whole blood will be recorded.
Changes from baseline in PT of Laboratory Examination | within 180 days after administration
  Prothrombin time (PT) is a screening test for exogenous coagulation factors
Changes from baseline in INR of Laboratory Examination | within 180 days after administration
  International standardized ratio (INR) is calculated from prothrombin time and international sensitivity index (ISI) of the reagent.
Changes from baseline in APTT of Laboratory Examination | within 180 days after administration
  Activated partial thromboplastin time (APTT) is a screening test for endogenous coagulation factors
Changes from baseline in total bilirubin of Laboratory Examination | within 180 days after administration
  Changes of total bilirubin concentration (μmol/L) in serum will be recorded
Changes from baseline in direct bilirubin of Laboratory Examination | within 180 days after administration
  Changes of direct bilirubin concentration (μmol/L) in serum will be recorded
Changes from baseline in ALT of Laboratory Examination | within 180 days after administration
  Changes of ALT concentration (U/L) in serum will be recorded
Changes from baseline in AST of Laboratory Examination | within 180 days after administration
  Changes of AST concentration (U/L) in serum will be recorded
Changes from baseline in total protein of Laboratory Examination | within 180 days after administration
  Changes of total protein concentration (g/L) in serum will be recorded
Changes from baseline in albumin of Laboratory Examination | within 180 days after administration
  Changes of albumin concentration (g/L) in serum will be recorded
Changes from baseline in total bile acid of Laboratory Examination | within 180 days after administration
  Changes of total bile acid concentration (μmol/L) in serum will be recorded
Changes from baseline in urea of Laboratory Examination | within 180 days after administration
  Changes of urea concentration (mmol/L) in serum will be recorded
Changes from baseline in creatinine of Laboratory Examination | within 180 days after administration
  Changes of creatinine concentration (μmol/L) in serum will be recorded
Changes from baseline in uric acid of Laboratory Examination | within 180 days after administration
  Changes of uric acid concentration (μmol/L) in serum will be recorded
Changes from baseline in glucose of Laboratory Examination | within 180 days after administration
  Changes of glucose concentration (mmol/L) in serum will be recorded
Changes from baseline in potassium of Laboratory Examination | within 180 days after administration
  Changes of potassium concentration (mmol/L) in serum will be recorded
Changes from baseline in sodium of Laboratory Examination | within 180 days after administration
  Changes of sodium concentration (mmol/L) in serum will be recorded
Changes from baseline in chlorine of Laboratory Examination | within 180 days after administration
  Changes of chlorine concentration (mmol/L) in serum will be recorded
Changes from baseline in Detection of infectious diseases of Laboratory Examination | within 180 days after administration
  It refers to infectious diseases screening
Changes from baseline in IgA of Laboratory Examination | within 180 days after administration
  Changes of IgA concentration （g/L）in serum will be recorded
Changes from baseline in IgG of Laboratory Examination | within 180 days after administration
  Changes of IgG concentration （g/L）in serum will be recorded
Changes from baseline in IgM of Laboratory Examination | within 180 days after administration
  Changes of IgM concentration （g/L）in serum will be recorded
Changes from baseline in total IgE of Laboratory Examination | within 180 days after administration
  Changes of total IgE concentration （g/L）in serum will be recorded
Changes from baseline in Pregnancy test of Laboratory Examination | within 180 days after administration
  Pregnancy test will be tested in female subjects
Changes from baseline in urine specific gravity of Laboratory Examination | within 180 days after administration
  Changes of urine specific gravity will be recorded
Changes from baseline in urine pH of Laboratory Examination | within 180 days after administration
  Changes of urine pH value will be recorded
Changes from baseline in urine glucose of Laboratory Examination | within 180 days after administration
  Changes of urine glucose will be examined by qualitative test (positive or negative)
Changes from baseline in urine protein of Laboratory Examination | within 180 days after administration
  Changes of urine protein will be examined by qualitative test (positive or negative)
Changes from baseline in urine ketone body of Laboratory Examination | within 180 days after administration
  Changes of urine ketone body will be examined by qualitative test (positive or negative)
Changes from baseline in urine white blood cell of Laboratory Examination | within 180 days after administration
  Changes of white blood cell in urine will be examined by qualitative test (positive or negative)
Changes from baseline in urine bilirubin of Laboratory Examination | within 180 days after administration
  Changes of urine bilirubin will be examined by qualitative test (positive or negative)
Changes from baseline in urine occult blood of Laboratory Examination | within 180 days after administration
  Changes of urine occult blood will be examined by qualitative test (positive or negative)
Changes from baseline in ECG PR interval | within 180 days after administration
  The cardiac rhythm is showed in 12 Leads Ambulatory Electrocardiogram in the form of continuous curve. Changes of this continuous curve will be recorded.
Changes from baseline in ECG QRS interval | within 180 days after administration
  The cardiac rhythm is showed in 12 Leads Ambulatory Electrocardiogram in the form of continuous curve. Changes of this continuous curve will be recorded.
Changes from baseline in ECG RR interval | within 180 days after administration
  The cardiac rhythm is showed in 12 Leads Ambulatory Electrocardiogram in the form of continuous curve. Changes of this continuous curve will be recorded.
Changes from baseline in ECG QT interval | within 180 days after administration
  The cardiac rhythm is showed in 12 Leads Ambulatory Electrocardiogram in the form of continuous curve. Changes of this continuous curve will be recorded.
Incidence of Treatment-Emergent Adverse Event | within 180 days after administration
  Incidence of Treatment-Emergent Adverse Events and Serious Adverse Events during the study period, and the severity of adverse events is determined according to the NCI CTCAE version 5.0
Change from baseline in Clinical Attachment Level (AL) | at baseline, 90 days, 180 days
  Clinical Attachment Level (AL) may be assessed to the nearest millimeter by means of a graduated probe and expressed as the distance in millimeters from the CEJ to the bottom of the probeable gingival/periodontal pocket
Change from baseline in Tooth Mobility (TM) | at baseline, 90 days, 180 days
  The continuous loss of the supporting tissues during periodontal disease progression may result in increased tooth mobility, which is divided into 3 degree: I°, II°, and III°. Changes from baseline in tooth mobility will be recorded
Change from baseline in Probing Depth (PD) | at baseline, 90 days, 180 days
  The probing depth is the distance from the gingival margin to the bottom of the gingival sulcus/pocket, is measured to the nearest millimeter by means of periodontal probe
Change from baseline in Gingival recession （GR） | at baseline, 90 days, 180 days
  Exposure of the tooth through apical migration of the gingiva is called gingival recession. Recorded as the distance in millimeters from the CEJ to the gingival margin
Change from baseline in Probing bleeding on probing (BOP) | at baseline, 90 days, 180 days
  A periodontal probe is inserted to the "bottom" of the gingival/periodontal pocket applying light force and is moved gently along the tooth (root) surface. If bleeding is provoked by this examination, the site examined is considered bleeding on probing-positive and, hence, inflamed. Probing Bleeding Index is divided into 5 grades: 0, 1, 2, 3 and 4.

OTHER OUTCOMES:
Change from baseline in interleukin-6 (IL-6) | at baseline, 90 days, 180 days，360 days，720 days
  Changes in IL-6 baseline will be confirmed through gingival crevicular fluid detection at D90 D180 D360 and D720
Change from baseline in tumor necrosis factor-alpha (TNF-α) | at baseline, 90 days, 180 days，360 days，720 days
  Changes in TNF-α baseline will be confirmed through gingival crevicular fluid detection at D90 D180 D360 and D720
Change from baseline in matrix metalloproteinase-8 (MMP-8) | at baseline, 90 days, 180 days，360 days，720 days
  Changes in MMP-8 baseline will be confirmed through gingival crevicular fluid detection at D90 D180 D360 and D720
Change from baseline in interleukin-1beta (IL-1β) | at baseline, 90 days, 180 days，360 days，720 days
  Changes in IL-1β baseline will be confirmed through gingival crevicular fluid detection at D90 D180 D360 and D720
Change from baseline in osteoprotegerin (OPG) | at baseline, 90 days, 180 days，360 days，720 days
  Changes in OPG baseline will be confirmed through gingival crevicular fluid detection at D90 D180 D360 and D720
Changes from baseline in height of the periodontal bone defect | at baseline, 360 days，720 days
  Changes from baseline in height of the periodontal bone defect which will be examined by CBCT at D360 and D720
Change from baseline in Clinical Attachment Level (AL) | at baseline, 360 days，720 days
  Clinical Attachment Level (AL) may be assessed to the nearest millimeter by means of a graduated probe and expressed as the distance in millimeters from the CEJ to the bottom of the probeable gingival/periodontal pocket
Change from baseline in Probing Depth (PD) | at baseline, 360 days，720 days
  The probing depth is the distance from the gingival margin to the bottom of the gingival sulcus/pocket, is measured to the nearest millimeter by means of periodontal probe
Change from baseline in Tooth Mobility (TM) | at baseline, 360 days，720 days
  The continuous loss of the supporting tissues during periodontal disease progression may result in increased tooth mobility, which is divided into 3 degree: I°, II°, and III°. Changes from baseline in tooth mobility will be recorded
Change from baseline in Gingival recession （GR） | at baseline, 360 days，720 days
  Exposure of the tooth through apical migration of the gingiva is called gingival recession. Recorded as the distance in millimeters from the CEJ to the gingival margin
Change from baseline in Probing bleeding on probing (BOP) | at baseline, 360 days，720 days
  A periodontal probe is inserted to the "bottom" of the gingival/periodontal pocket applying light force and is moved gently along the tooth (root) surface. If bleeding is provoked by this examination, the site examined is considered bleeding on probing-positive and, hence, inflamed. Probing Bleeding Index is divided into 5 grades: 0, 1, 2, 3 and 4.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Wang, Master, Principal Investigator — Department of Stomatology, Peking University Third Hospital, Beijing, China
Locations (1):
- Peking University Third Hospital, Beijing, Beijng, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Y, Liu Y, Hu J, Han J, Song L, Liu X, Han N, Xia X, He J, Meng H, Wan M, Wang H, Liu X, Gao Z, Wang X, Wu C, Wang S. Impact of allogeneic dental pulp stem cell injection on tissue regeneration in periodontitis: a multicenter randomized clinical trial. Signal Transduct Target Ther. 2025 Jul 31;10(1):239. doi: 10.1038/s41392-025-02320-w. PMID 40739139